CLINICAL TRIAL: NCT06513065
Title: A Single Blinded Randomised Controlled Study to Evaluate the Non-inferiority of HIPEC with Mitomycin C 10 Mg/m2 for 60 Minutes Versus HIPEC with Mitomycin C 35mg/m2 for 90 Minutes in the Treatment of Pseudomyxoma Peritonei from Perforated Epithelial Mucinous Tumours of the Appendix
Brief Title: Study to Evaluate the Non-inferiority of Low-dose HIPEC Versus High-dose HIPEC in the Treatment of PMP (HIPEC-PMP)
Acronym: HIPEC-PMP
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Southampton (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 83709
Record Dates: First submitted 2024-06-25; First posted 2024-07-22 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-07

CONDITIONS: Pseudomyxoma Peritonei
Keywords: Psuedomyxoma Peritonei; Mitomycin C; Hyperthermic Intraperitoneal Chemotherapy; Appendix
MeSH Terms: conditions — Pseudomyxoma Peritonei | interventions — Mitomycin; Hyperthermic Intraperitoneal Chemotherapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ARM A (lower dose) (Active Comparator): 10mg/m2 MMC given intraperitoneal as one single dose at Time 0 of HIPEC
  Interventions: Drug: Mitomycin c
- ARM B (higher dose) (Experimental): 35mg/m2 MMC given in fractionated doses :50% at Time 0, 25% at T30 and 25% at T60
  Interventions: Drug: Mitomycin c

INTERVENTIONS:
Drug: Mitomycin c — Mitomycin is a tumour antibiotic isolated from the broth of Streptomyces species. It has alkylating properties, which results in DNA cross-linking. Once MMC enters the tumour cell, it needs microsomal modification by various enzymes to be transformed into active state; free radicals constituted of semiquinones of MMC are responsible for its cytotoxic effects.
  Mitomycin is licenced in the UK and recommended by NICE for intraperitoneal chemotherapy.
  Other Names: HIPEC

SUMMARY:
The Investigators are researching how to improve the treatment currently available for patients diagnosed with Pseudomyxoma Peritonei (PMP). This is a rare cancer that usually starts in the appendix and spreads around the abdomen.

PMP is usually treated using a type of surgery called Cytoreductive Surgery (CRS). During the surgery heated chemotherapy will also be used to treat any cancer cells that cannot be seen and may be left behind. This is called Hyperthermic Intraperitoneal Chemotherapy (HIPEC).

This treatment is commonly used in the UK and in Europe, however, the chemotherapy can be given at two different doses: a lower dose over 60 minutes or a higher-dose over 90 minutes.

The Investigators want to understand if there is a difference between these two doses. The higher dose has been associated with a slightly increased rate of complications but may be better at killing cancer cells and preventing recurrence of cancer. In Basingstoke the lower dose over 60 minutes is used and survival results are similar to centres who use the higher dose.

Previous studies have shown that both doses are effective at treating PMP, but no research has shown which is better for patients. The Investigators hope to show that the lower-dose over 60-minutes is as good as the higher-dose over 90-minutes.

DETAILED DESCRIPTION:
HIPEC-PMP is a randomised, non-inferiority phase III trial with two parallel groups, designed to assess two doses of mitomycin C (MMC) for the treatment of pseudomyxoma peritonei. The trial is to be carried out in a single specialist centre.

The low and high doses within the trial are used routinely across the world, but to date they have not been compared directly. As the lead site use low dose MMC, the trial has been designed to assess whether this has comparable performance to high dose with respect to clinical outcomes (primarily disease-free survival; DFS), hence the non-inferiority design. The trial uses a Bayesian design to incorporate existing information on the two treatments (given they are used routinely, and various studies have reported DFS rates in cohort studies). The design allows for discounting the prior information through data-driven weighting of different prior distributions, if the observed data is observed to be markedly different to prior data.

Cytoreductive surgery (CRS) and hyperthermic intraperitoneal chemotherapy (HIPEC) represent the standard of care for Pseudomyxoma Peritonei (PMP) of appendiceal origin. Although Mitomycin C is used as standard of care HIPEC treatment, the optimal dose of Mitomycin C (MMC) and duration of HIPEC following cytoreductive surgery remains to be defined.

This study therefore aims to evaluate the non-inferiority of HIPEC with mitomycin C 10 mg/m2 for 60 minutes versus HIEPC with mitomycin C 35 mg/m2 for 90 minutes. There is a small risk of higher toxicity with 35 mg/m2 of Mitomycin C, however Kuijpers et al found that morbidity was tolerable and convincing survival.

There is limited evidence on the quality of life in patients with PMP, therefore assessing quality of life will provide information that could be used to improve patient care and well-being. In addition, furthering understanding of the genetics of the disease could improve prognostication and targeted treatments for patient benefit could be explored and will therefore be investigated in this study. Translational blood samples including tissue (normal, primary and metastatic), serum, plasma, DNA, RNA and buffy coat will be collected for genetic analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical and/or radiological diagnosis of pseudomyxoma peritonei from a primary mucinous epithelial tumours of the appendix (low and high grade)
2. The extent of intraperitoneal disease must be deemed to be amenable to complete cytoreduction (CC0-1, i.e. residual disease of < 2.5mm in diameter).
3. Patients aged 16 or more and capable of giving informed consent for the procedures and interventions of the current trial.
4. ECOG performance status 0-1.

   Exclusion Criteria:
5. Patients who have previously undergone cytoreductive surgery and/or intraperitoneal chemotherapy.
6. Clinical evidence or suspicion of metastases to sites different than peritoneum or intra-abdominal lymph nodes
7. Hypersensitivity to the active substance (mitomycin) or its excipients (mannitol, hydrochloric acid, sodium hydroxide)
8. Patients with conditions which may affect their ability to understand, retain and weigh up the information related to the requirements and consenting process of the study
9. Women who are pregnant or breastfeeding.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2024-12-04 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Disease Free Survival | 24 Months
  To compare disease free survival between low- and high-dose mitomycin C (MMC).

SECONDARY OUTCOMES:
Adverse Events using Common Terminology Criteria for Adverse Events | 24 Months
  To compare short- and long-term toxicity between arms.
EQ-5D-5L Quality of Life Questionnaire | 24 Months
  To compare short- and long-term quality of life between arms.
QLQ-C30 Quality of Life Questionnaire | 24 Months
  To compare short- and long-term quality of life between arms.
MODRUM Healthcare Resource Use Questionnaire | 24 Months
  To compare the cost-effectiveness of high dose with low dose mitomycin. Participants will document how often they have used healthcare services over a period of 2 years following surgery. The number of uses of healthcare services reported by participants will be compared between the two arms.
Healthcare Cost | 24 Months
  To compare the cost-effectiveness of high dose with low dose mitomycin. Participants will document how often they have used healthcare services over a period of 2 years following surgery using the MODRUM questionnaire. The number of reported uses of healthcare services and associated costs of using these services will be compared between the two arms.
Quality-adjusted Life Years | 24 Months
  Results from the EQ-5D-5L Quality of Life Questionnaire, QLQ-C30 Quality of Life Questionnaire, and MODRUM Healthcare Resource Use Questionnaire as reported by participants will be used to calculate quality-adjusted life years for participants. The results will be compared between the two arms.

CONTACTS AND LOCATIONS:
Overall Officials: Faheez Mohamed, MBChB, MD, FRCS, Principal Investigator — Peritoneal Malignancy Unit Hampshire Hospitals NHS Foundation Trust
Locations (1):
- Peritoneal Malignancy Institute Basingstoke - Hampshire Hospitals NHS Foundation Trust, Basingstoke, Hampshire, United Kingdom